CLINICAL TRIAL: NCT03645304
Title: Postoperative Analgesic Efficacy of Continuous Wound Infusion With Local Anesthetics After Laparoscopy (PAIN): a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Postoperative Analgesic Efficacy of Continuous Wound Infusion After Laparoscopy
Acronym: PAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-05-014
Record Dates: First submitted 2018-05-03; First posted 2018-08-24 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Benign Gynecologic Neoplasm
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine group (Experimental): Continuous wound infusion device used in this study was ON-Q Painbuster Silver Soaker (I-Flow Corporation, Lake Forest, CA, USA) comprised an elastomeric pump maintaining constant pressure to infuse 2ml/hour of analgesic to the wound through a catheter for 50 hours. In all participants, the surgeon inserted a 20-gauge, 6.5-cm, multi-holed soaker catheter through an introducer needle after closure of the transumbilical fascia. The catheter was located in the deep subcutaneous space, above the fascia near the skin incision. In the experimental group, an elastomeric pump filled with local analgesic solution (total volume 100ml) containing 750mg ropivacaine .
  Interventions: Drug: Ropivacaine; Device: ON-Q Painbuster Silver Soaker
- 0.9% Saline group (Placebo Comparator): Continuous wound infusion device used in this study was ON-Q Painbuster Silver Soaker (I-Flow Corporation, Lake Forest, CA, USA) comprised an elastomeric pump maintaining constant pressure to infuse 2ml/hour of analgesic to the wound through a catheter for 50 hours. In all participants, the surgeon inserted a 20-gauge, 6.5-cm, multi-holed soaker catheter through an introducer needle after closure of the transumbilical fascia. The catheter was located in the deep subcutaneous space, above the fascia near the skin incision. In the control group, an elastomeric pump filled with filled with 100ml of 0.9% saline .
  Interventions: Drug: 0.9% saline group

INTERVENTIONS:
Drug: Ropivacaine — Continuous wound infusion device used in this study was ON-Q Painbuster Silver Soaker (I-Flow Corporation, Lake Forest, CA, USA) comprised an elastomeric pump maintaining constant pressure to infuse 2ml/hour of analgesic to the wound through a catheter for 50 hours. In all participants, the surgeon inserted a 20-gauge, 6.5-cm, multi-holed soaker catheter through an introducer needle after closure of the transumbilical fascia. The catheter was located in the deep subcutaneous space, above the fascia near the skin incision. In the experimental group, an elastomeric pump filled with local analgesic solution (total volume 100ml) containing 750mg ropivacaine .
  Ropivacaine is local analgesics.
  Arms: Ropivacaine group
Drug: 0.9% saline group — Continuous wound infusion device used in this study was ON-Q Painbuster Silver Soaker (I-Flow Corporation, Lake Forest, CA, USA) comprised an elastomeric pump maintaining constant pressure to infuse 2ml/hour of analgesic to the wound through a catheter for 50 hours. In all participants, the surgeon inserted a 20-gauge, 6.5-cm, multi-holed soaker catheter through an introducer needle after closure of the transumbilical fascia. The catheter was located in the deep subcutaneous space, above the fascia near the skin incision. In the control group, an elastomeric pump filled with filled with 100ml of 0.9% saline .
  Arms: 0.9% Saline group
Device: ON-Q Painbuster Silver Soaker — ON-Q Painbuster Silver Soaker (I-Flow Corporation, Lake Forest, CA, USA)
  Arms: Ropivacaine group

SUMMARY:
Studies evaluating the effectiveness of continuous wound infusion (CWI) to manage postoperative pain following laparoscopy are markedly lacking. Especially, there was no study comparing CWI and placebo in treating gynecologic laparoscopy. Therefore, the investigators conducted this randomized, double-blind, placebo-controlled trial to investigate whether CWI of local anesthetics was an effective strategy for enhanced recovery after surgery (ERAS), compared with placebo in patients undergoing benign gynecologic laparoscopy.

DETAILED DESCRIPTION:
Laparoscopic surgery has become an acceptable alternative for open surgery in treating benign gynecologic diseases. One of most important advantages of laparoscopy is a reduced postoperative pain compared with open surgery. Moreover, postoperative pain plays an important part in the enhanced recovery after surgery (ERAS) pathway. Although the length of hospitalization and recovery period after laparoscopy tends to be shorter, postoperative pain can still be an important issue.

Recently, continuous wound infusion (CWI) providing a constant flow of local anesthetic directly a surgical wound postoperatively has been widely used to reduce pain after cesarean section and open surgery. Studies evaluating the effectiveness of CWI to manage postoperative pain following laparoscopy are markedly lacking. Especially, there was no study comparing CWI and placebo in treating gynecologic laparoscopy. Therefore, the investigators conducted this randomized, double-blind, placebo-controlled trial to investigate whether CWI of local anesthetics was an effective strategy for ERAS, compared with placebo in patients undergoing benign gynecologic laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years,
* American Society of Anesthesiologists physical status (ASAPS) classification I-II
* the absence of pregnancy at the time of surgery

Exclusion Criteria:

* allergy to amide local anesthetics including ropivacaine
* laparoscopic surgery needing ≥ 3 separate skin incisions
* history of ventral or incisional hernia
* pre-existing coagulopathy, neurologic or cognitive dysfunction
* systemic or regional (especially, umbilicus) infection
* previously taking opioids for acute or chronic pain
* inability to accurately express their pain.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-04-03 (Estimated); Study Completion 2020-04-03 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 24-hour after surgery
  The postoperative pain was measured using a visual analog scale (VAS) at 24 hours after surgery by several assessors who were blinded to the interventions. The scale was presented as a 10-cm line with verbal descriptors ranging from "no pain" to "worst imaginable pain".

SECONDARY OUTCOMES:
the number of rescue analgesics | within 3days after surgery
  Rescue analgesia (75 mg diclofenac sodium administered intramuscularly or 25mg pethidine intramuscularly) was provided upon participant request

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital, Seoul, Republic of Korea
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No